CLINICAL TRIAL: NCT04587245
Title: The Provider Insurance Revenue Study
Brief Title: The Provider Insurance Revenue Study in Healthcare Providers in the United States of America
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: ND Sciences, LLC (Industry)
Collaborators: University of California, Irvine (Other)
Responsible Party: Sponsor
Other Study IDs: PIRStudy
Record Dates: First submitted 2020-10-07; First posted 2020-10-14 (Actual); Last update posted 2021-10-18 (Actual); Status verified 2021-10

CONDITIONS: Covid19; Financial Disclosure
Keywords: Healthcare providers; Covid19; Financial impact; Income
MeSH Terms: conditions — COVID-19 | interventions — Interviews as Topic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Physicians: Physician or healthcare Provider based anywhere in the United States who is eligible to submit claims to an insurance company on behalf of patients
  Interventions: Other: Online questionnaire and interviews

INTERVENTIONS:
Other: Online questionnaire and interviews — Online questionnaire, financial statements (one month per quarter in 2020) submitted electronically, interview with professional accounting firm and review of data and exit Interview

SUMMARY:
The investigators are enrolling 100 healthcare Provider volunteers (n=100) from across the United States to help to evaluate and document the financial impact of COVID-19 on Physicians and other healthcare Providers. This investigation will compare individual Physician revenues before and after the advent of the COVID-19 pandemic. The investigators expect to be able to differentiate between revenues lost due to the COVID-19-driven business recession and revenues lost due to the manipulation of reimbursement processes by insurance companies. The inextricable linkage between Payer and Physician revenues suggests that Payer revenues are higher at the direct expense of Physicians, since both streams come from the same sources of funding. The secondary objective is aimed at revealing the methods Payers use to retain more money.

DETAILED DESCRIPTION:
Since the beginning of the COVID-19 pandemic in March, 2020, Physicians and other medical Providers have taken devastating hits to their practice revenues. Most of the losses are due to doctors being forced to curtail elective procedures and office visits as Americans were ordered to stay home during the height of the national health emergency.

As Physicians were able to return to work in the early Summer, even if only partially, many had to adjust to the newer medical practice of telehealth, and the lower revenues that came with it. The Centers for Medicare & Medicaid Services (CMS) gave assurances to Physicians that Medicare would reimburse telehealth encounters at 100% of the office visit rate. But private Payers were under no such obligation. Across the country, Physicians are reporting that they're being reimbursed at about 70% of an office visit rate despite the fact that telehealth requires both resources and expertise to implement effectively, and each encounter takes up to twice as long as an office visit.

Adding to financial hardships, Physicians across the nation are reporting that legitimate insurance claims are being held up and denied by the insurance companies at a higher rate than ever, cutting off the cash that they need so desperately. As of June 1, only half of Physician practices say they have enough cash to stay open for another month.

In just 2 months in the spring of 2020, over 45 million Americans lost their jobs and for many, that also meant the loss of their employment-related health insurance. Despite shedding a massive number of members from their rolls, health insurance companies are actually predicting record profits for 2020. The pandemic it seems, is very good indeed for the health insurance business. Private investors and executives are taking huge dividends and bonuses out of the system just at a time when US healthcare needs a vast new investment of healthcare resources into the system. The good fortune of a few individuals and corporations comes at an as yet untold expense to American society.

The formula for insurance company success in a pandemic only happens one way. By keeping member premiums, delaying payments, and denying treatment authorizations, the large health insurance companies are taking advantage of the profound misfortunes of both doctors and patients during a national health emergency.

The COVID-19 pandemic will have adverse effects on the health of Americans that will be sprawling and long-felt. However, it is not for this study to decide whether private interests will always be antithetical to public interests when it comes to healthcare. That is a public debate that will continue to evolve as the profound weaknesses of the American way of distributing healthcare are magnified and exposed in a time of social upheaval.

The investigators do know that in order to get a handle on the major damage we see occurring in real-time- and to inform that debate, it is first necessary to measure it.

ELIGIBILITY:
Inclusion Criteria:

* Healthcare Provider based anywhere in the United States who is eligible to submit claims to an insurance company on behalf of patients.
* To agree to participate in this study

Exclusion Criteria:

* Any condition that at the discretion of the principal investigator renders the subject ineligible to participate in this study.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Healthcare Provider based anywhere in the United States who is eligible to submit claims to an insurance company on behalf of patients.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-10-01 (Actual); Primary Completion 2022-10-15 (Estimated); Study Completion 2022-10-15 (Estimated)

PRIMARY OUTCOMES:
Change in monthly income of healthcare Providers from baseline to 6, 9 and 12 months after the beginning of the COVID-related events | 12 months
  Change in monthly income of healthcare Providers from baseline to 6, 9 and 12 months after the beginning of the COVID-related events

SECONDARY OUTCOMES:
Differences in Accounts Receivable (AR) due to claim denials over 4 quarters: Differences in recoveries of AR. | 12 months
  Differences in Accounts Receivable (AR) due to claim denials over 4 quarters: Differences in recoveries of AR.

CONTACTS AND LOCATIONS:
Overall Officials: Henry Broeska, PhD, Principal Investigator — University of California Irvine Beall Applied Innovation
Locations (1):
- University of California Irvine Beall Applied Innovation, Irvine, California, United States

IPD SHARING:
Plan to Share IPD: No